CLINICAL TRIAL: NCT01510561
Title: A Ph Ib Study of Fractionated 90Y-hPAM4 Plus Gemcitabine in Pancreatic Cancer Patients Receiving at Least 2 Prior Therapies.
Brief Title: A Study of Fractionated 90Y-hPAM4 Plus Gemcitabine in Pancreatic Cancer Patients Receiving at Least 2 Prior Therapies.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no subjects enrolled
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hPAM4-03
Record Dates: First submitted 2012-01-05; First posted 2012-01-16 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: metastatic pancreatic adenocarcinoma; pancreatic cancer; metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — clivatuzumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 90Y-hPAM4 (Experimental): 90Y-hPAM4 is administered weekly for 3 weeks
  Interventions: Drug: 90Y-hPAM4
- 90Y-hPAM4 + gemcitabine (Experimental): 90Y-hPAM4 is administered weekly for 3 weeks, while gemcitabine is administered weekly for 4 weeks.
  Interventions: Drug: 90Y-hPAM4; Drug: 90Y-hPAM4 + gemcitabine

INTERVENTIONS:
Drug: 90Y-hPAM4 — 90Y-hPAM4 will be administered weekly for 3 weeks in conjunction with gemcitabine which will be administered weekly x 4.
  Other Names: Clivatuzumab Tetraxetan
Drug: 90Y-hPAM4
  Other Names: clivatuzumab tetraxetan
Drug: 90Y-hPAM4 + gemcitabine
  Other Names: gemzar; clivatuzumab tetraxetan
  Arms: 90Y-hPAM4 + gemcitabine

SUMMARY:
90Y-hPAM4 is administered weekly for 3 weeks combined with 4 weekly doses of gemcitabine to assess. This is a dose escalation study of 90Y-hPAM4 to assess which dose is safe and effective as 3rd line treatment for patients with metastatic pancreatic cancer. Patients are then followed weekly for 12 weeks and afterwards for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ≥ 18 years of age, who are able to understand and give written informed consent
* Histologically or cytologically confirmed pancreatic adenocarcinoma
* Stage IV (metastatic) disease, including patients who underwent surgery but had incomplete resections
* Previously treated and received two prior treatment regimens for advanced disease
* Karnofsky performance status ≥ 60 % (Appendix A)
* Expected survival ≥ 3 months
* At least 4 weeks beyond major surgery, 2 weeks beyond chemotherapy, radiotherapy, other experimental treatments
* At least 2 weeks beyond corticosteroids, except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, ANC > 1,500 per mm3, platelets > 100,000 per mm3)
* Adequate renal and hepatic function (creatinine and bilirubin ≤ 1.5 X IULN, AST and ALT ≤ 2.0 X IULN [5.0 X IULN if due to liver metastases])
* Otherwise, all toxicity at study entry ≤ Grade 1 by NCI CTC v3.0 or recovered to baseline or discussed with and agreed to with Immunomedics' Medical Monitor.

Exclusion Criteria:

* Women who are pregnant or lactating
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period
* Known metastatic disease to the central nervous system
* Presence of bulky disease (defined as any single mass > 10 cm in its greatest dimension)
* Patients with > Grade 2 nausea or vomiting and/or signs of intestinal obstruction
* Prior radiation dose > 3,000 cGy to the liver, > 2,000 cGy to lungs and kidneys or prior external beam irradiation to a field that includes more than 30% of the red marrow
* Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least a 3-year disease free interval
* Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive
* Known history of active coronary artery disease, unstable angina, myocardial infarction, or congestive heart failure present within 6 months, or cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy
* Known history of active COPD, or other moderate-to-severe respiratory illness present within 6 months
* Known autoimmune disease or presence of autoimmune phenomena (except rheumatoid arthritis requiring only low dose maintenance corticosteroids)
* Infection requiring intravenous antibiotic use within 1 week
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety (change in hematology and chemistry laboratory values from baseline) | 1 year
  Acute safety will be assessed weekly for the 1st 12 weeks, and then for up to 1 year after completion of study drug treatment. Safety will be assessed by comparing baseline hematology and chemistry laboratory values with the values obtained weekly after treatment. Safety will also be assessed by the adverse events that are reported.

SECONDARY OUTCOMES:
Dosage determination | 2 years
  This study is also being done to determine an acceptable 90Y-hPAM4 dose in this patient population. It is anticipated that enrollment will occur over 2 years.
Efficacy | 1 year
  Efficacy will be assessed for at least 1 year after treatment with study drug. CT scans will be used to determine treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: William A Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (24):
- United States (24):
  - Banner Healthcare, Gilbert, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Christiana Care Health Services Helen Graham Cancer Center, Newark, Delaware
  - Sylvester Comprehensive Cancer Center Univ. Miami, Miami, Florida
  - Jackson North Medical Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Mountain States Tumor Institute, Boise, Idaho
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Detroit Clinical Research Center, Detroit, Michigan
  - St. Mary's Trinity Healthcare, Grand Rapids, Michigan
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Weill Cornell NY Presbyterian Hospital, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Kimmel Cancer Center at Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Institute of Translational Oncology Research, Greenville, South Carolina
  - Tyler Cancer Center, Tyler, Texas
  - VA Oncology Associates, Norfolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Picozzi VJ, Ramanathan RK, Lowery MA, Ocean AJ, Mitchel EP, O'Neil BH, Guarino MJ, Conkling PR, Cohen SJ, Bahary N, Frank RC, Dragovich T, Bridges BB, Braiteh FS, Starodub AN, Lee FC, Gribbin TE, Richards DA, Lee M, Korn RL, Pandit-Taskar N, Goldsmith SJ, Intenzo CM, Sheikh A, Manzone TC, Horne H, Sharkey RM, Wegener WA, O'Reilly EM, Goldenberg DM, Von Hoff DD. (90)Y-clivatuzumab tetraxetan with or without low-dose gemcitabine: A phase Ib study in patients with metastatic pancreatic cancer after two or more prior therapies. Eur J Cancer. 2015 Sep;51(14):1857-64. doi: 10.1016/j.ejca.2015.06.119. Epub 2015 Jul 14. PMID 26187510